CLINICAL TRIAL: NCT00905788
Title: Embryo Transfer: Embryo Expulsion and Outcome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi, Chief, Royan Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-001
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Infertility
Keywords: Embryo transfer; IVF/ICSI; Embryo expulsion
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Embryo transfer without any intervention
- Embryo Expulsion (Experimental)
  Interventions: Procedure: prevention of embryo expulsion

INTERVENTIONS:
Procedure: prevention of embryo expulsion — The prevention of embryo expulsion will be carried out after embryo transfer
  Arms: Embryo Expulsion

SUMMARY:
According to the studies, about 80% of patients undergoing in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) reach to the embryo transfer process, but only a few of them become pregnant.

The cause of this difference can be due to some factors such as the endometrial receptivity, quality of transferred embryos and embryo transfer technique. Retained or expelled embryo(s) following embryo transfer is (are) one of the factors which may be effective on outcome. The purpose of this randomized clinical trial study is "Lowering embryo expulsion following embryo transfer to improve outcome."

DETAILED DESCRIPTION:
A total of 134 infertile women who undergo IVF or ICSI treatment cycle at Royan Institute (Infertility and Reproductive Medicine Research Centre) will enroll in this prospective randomized clinical trial study and will randomly be divided into two groups of 67 patients. This study has been approved by Royan ethics committee and written consent will be obtained from each patient. The patients with frozen-thawed embryo transfer cycle and those with oocyte donation cycle, the women with uterine abnormality and the subjects with submucosal and intramural myoma, will be excluded from this study.

After the ovarian stimulation and oocyte retrieval, The IVF and intracytoplasmic sperm injection (ICSI) procedures will be performed to produce the embryos.

Embryo transfer will be done only by one skilled physician. The patients will be divided into two groups of A and B by computerized randomly chart. In group A, the prevention technique of embryo expulsion will be carried out following embryo transfer, but no intervention will be performed in group B (control group).

After 2 weeks, the patients will be tested for serum β-hCG for assessing the pregnancy. The clinical pregnancy will be clarified by the number of women with gestational sacs on transvaginal sonography at 4-6 weeks of gestation. In the calculation of implantation, the number of gestational sacs will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF or ICSI treatment cycle
* Patients with "long or antagonist" protocol

Exclusion Criteria:

* The patients with frozen-thawed embryo transfer cycle
* Those with oocyte donation cycle
* The women with uterine abnormality
* The women with submucosal and intramural myoma
* Who does not have good-quality embryos appropriate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 4-6 weeks

SECONDARY OUTCOMES:
Implantation rate | 6-7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tahere Madani, MD, Principal Investigator — Royan Institute; Mahnaz Ashrafi, MD, Principal Investigator — Royan Institute
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- See also: Official site — http://www.royaninstitute.org